CLINICAL TRIAL: NCT03508414
Title: Nutritional Approaches in Multiple Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Friedemann Paul, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: NAMS-study
Record Dates: First submitted 2017-12-21; First posted 2018-04-25 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis
Keywords: Relapse-remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ketogenic diet (Experimental)
  Interventions: Behavioral: ketogenic diet
- Intermittent therapeutical fasting (Experimental)
  Interventions: Behavioral: Intermittent therapeutical fasting
- Control group (Active Comparator): The control group is receiving a vegetarian-focused diet according to the current recommendations of the German Society for Nutrition (DGE) for MS patients.
  Interventions: Behavioral: Active comparator

INTERVENTIONS:
Behavioral: ketogenic diet — Patients receive a ketogenic diet, which is carbohydrate-reduced with a high amount of fat.
  Arms: Ketogenic diet
Behavioral: Intermittent therapeutical fasting — Patients fast for 1 week every six months. Additionally, the patients do an intermittent fasting, that is to say they do not eat for at least 14 hours a day.
  Arms: Intermittent therapeutical fasting
Behavioral: Active comparator — The control group is receiving a vegetarian-focused diet according to the current recommendations of the German Society for Nutrition (DGE) for MS patients.
  Arms: Control group

SUMMARY:
The aim of this project is to characterize the influence of a ketogenic diet and intermittent therapeutical fasting on the course of the disease, as measured by T2-hyperintense cerebral lesions with magnetic resonance tomography (MRT) in patients with multiple sclerosis (RRMS). The investigators expect in both intervention groups fewer cerebral T2 lesions occurring after 18 months in comparison to the control group and as detectable by MRT. According to current recommendations of the German Society of Nutrition (DGE), the control group receives a vegetarian-focused, anti-inflammatory diet.

ELIGIBILITY:
Inclusion Criteria:

* Existing health insurance, so that in case of random findings these can also be clarified
* Patients with relapsed-remitting MS according to the MS diagnostic criteria according to McDonald 2010
* Age 18-65
* Consent ability and written consent
* BMI between 19 and 45 kg / m2
* EDSS <4.5
* Stable immunomodulatory therapy or no immunomodulatory therapy> 6 months before confinement
* In the last 2 years ≥ 1 relapse or within the last 2 years ≥ 1 new T2 lesions or ≥ 1 contrast-sensitive lesion in MRT
* Consent that possible random findings are reported

Exclusion Criteria:

* Initiation or modification of immunomodulatory therapy during the study
* Cortisone treatment in the last 30 days before enrollment
* Relapse in the last 30 days before enrollment
* Insulin-dependent diabetes mellitus (type I)
* Intake of Omega 3 fatty acids (DHA, EPA) - more than 1 g / day
* Significant cognitive impairment, clinically relevant or progressive disease (e.g., liver, kidney, cardiovascular system, respiratory tract, vascular system, brain, metabolism, thyroid) that could affect the course of the study
* Malignant disease
* Simultaneous participation in an interventional study or participation in an interventional study in the last two months before study inclusion
* Clinically relevant addiction or substance abuse disorder (defined as alcohol, drug and drug abuse)
* Nicotine consumption of > 5 cigarettes per day and no willingness to stop consumption during therapeutic fasting.
* Insufficient mental possibility of cooperation
* Eating disorder
* Kidney stones
* Known metabolic disorders (e.g., fatty acid oxidation disorders, ketolysis / ketogenesis or glucogenesis disorder, hyperinsulinism (e.g., nesidioblastoma), pyruvate carboxylase deficiency)
* Therapy with oral anticoagulants (e.g., Marcumar)
* Pregnancy and breast feeding period
* Suspected lack of compliance
* Performing of a diet for weight reduction
* Special diet for medical reasons
* Change of the body weight of more than 5 kg within one month before the start of the Intervention
* Medical, psychiatric or other conditions that restrict the patient's following abilities: to interpret the study information, to give informed consent, to adhere to the rules of the protocol, or to complete the study
* Contraindications to MRT examinations [persons with metallic implants (e.g., intracranial metal clips) and carriers of electronic devices (e.g., pacemaker) or persons with claustrophobia]

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in cerebral T2 lesions from Baseline at 18 months | Change from baseline at 18 months
  Number of new cerebral T2 lesions in MRT after 18 months compared to baseline MRT

SECONDARY OUTCOMES:
Change in neurological-functional disability: physical and cognitive function | Change from baseline at 9 and 18 months
  influence of the interventions on cognitive and physical disability progression using Multiple Sclerosis Functional Composite (MSFC)
Change in neurological-functional disability : physical function | Change from baseline at 9 and 18 months
  influence of the interventions on physical disability progression using Expanded Disability Status Score (EDSS). The EDSS is assessing the progress of disability in MS patients with a scale between 0-12 points, while 0 indicates no disability and 10 indicates death through MS.
annual relapse rate | 12 months
  relapse rate
progress of brain atrophy | Change from baseline at 18 months
  PBVC = percent brain volume change

CONTACTS AND LOCATIONS:
Overall Officials: Friedemann Paul, Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bahr LS, Bock M, Liebscher D, Bellmann-Strobl J, Franz L, Pruss A, Schumann D, Piper SK, Kessler CS, Steckhan N, Michalsen A, Paul F, Mahler A. Ketogenic diet and fasting diet as Nutritional Approaches in Multiple Sclerosis (NAMS): protocol of a randomized controlled study. Trials. 2020 Jan 2;21(1):3. doi: 10.1186/s13063-019-3928-9. PMID 31898518